CLINICAL TRIAL: NCT06157580
Title: Balance of Angiotensin II Receptors in Vessel Function After Preeclampsia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Anna Stanhewicz, PhD (Other)
Responsible Party: Sponsor-Investigator, Anna Stanhewicz, PhD, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 202309383
Record Dates: First submitted 2023-11-27; First posted 2023-12-06 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Preeclampsia
Keywords: postpartum; vascular
MeSH Terms: conditions — Pre-Eclampsia | interventions — compound 21; Angiotensin II

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- History of a preeclampsia (Other): Women who had preeclampsia in their most recent pregnancy
  Interventions: Drug: Compound 21; Drug: Angiotensin II
- History of a healthy pregnancy (Other): Women who had an uncomplicated pregnancy
  Interventions: Drug: Compound 21; Drug: Angiotensin II

INTERVENTIONS:
Drug: Compound 21 — differences in vasodilation to compound 21 in the skin between groups
Drug: Angiotensin II — differences in vasoconstriction to angiotensin II in the skin between groups

SUMMARY:
Otherwise healthy women who develop preeclampsia during pregnancy are more likely to develop and die of cardiovascular disease later in life. The reason why this occurs is unclear but may be related to impaired endothelial function and dysregulation of the angiotensin system that occurs during preeclampsia and persists postpartum, despite the remission of clinical symptoms. The purpose of this investigation is to determine the mechanisms contributing to this lasting blood vessel damage caused by reduced endothelial function in women who have had preeclampsia compared to women who had a healthy pregnancy. Identification of these mechanisms and treatment strategies may lead to better clinical management of cardiovascular disease risk in these women.

The purpose of this study is to examine differences in the microvascular balance of angiotensin II receptors women who have had preeclampsia. This will help the investigators better understand the mechanisms of dysregulated angiotensin II receptors in formerly preeclamptic women, and how activation or inhibition of these receptors may restore microvascular function.

In this study, the investigators use the blood vessels in the skin as a representative vascular bed for examining mechanisms of microvascular dysfunction in humans. Using a minimally invasive technique (intradermal microdialysis for the local delivery of pharmaceutical agents) the investigators examine the blood vessels in a dime-sized area of the skin.

ELIGIBILITY:
Inclusion Criteria:

* women who had preeclampsia and women who did not have preeclampsia
* 12 weeks to 5 years postpartum
* 18-45 years old

Exclusion Criteria:

* history of hypertension or metabolic disease before pregnancy
* history of gestational diabetes or gestational hypertension
* skin diseases
* current tobacco use
* current antihypertensive medication
* statin or other cholesterol-lowering medication
* currently pregnant or planning to become pregnant
* body mass index less than <18.5 or >30 kg/m2
* allergy to materials used during the experiment.(e.g. latex),
* known allergy to study drugs

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-12-08 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Change in microvascular angiotensin II (ang II) type 2 receptor (AT2R)-mediated dilation response measured by laser-Doppler flowmetry | at the study visit, an average of 4 hours
  cutaneous vascular vasodilator responses to compound 21 perfusion in lactated Ringer's and losartan treated microdialysis sites
Change in microvascular ang II-mediated constriction response measured by laser-Doppler flowmetry | at the study visit, an average of 4 hours
  cutaneous vascular vasoconstrictor responses to angiotensin II perfusion in lactated Ringer's and PD-123319 treated microdialysis sites

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No